CLINICAL TRIAL: NCT00497185
Title: Mindfulness-based Cognitive Therapy for Patients With Functional Disorders. A Randomized Controlled Trial
Brief Title: Mindfulness-based Cognitive Therapy for Patients With Functional Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: The Ministry of Science, Technology and Innovation, Denmark (Other Government); Aarhus University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 200706
Record Dates: First submitted 2007-07-04; First posted 2007-07-06 (Estimated); Last update posted 2011-11-16 (Estimated); Status verified 2011-11

CONDITIONS: Somatization Disorder; Functional Disorders; Bodily Distress Disorder
Keywords: Mindfulness-Based Cognitive Therapy; Somatization Disorder; Medically Unexplained Symptoms; Functional Somatic Symptoms; SF-36
MeSH Terms: conditions — Somatoform Disorders; Neurasthenia; Medically Unexplained Symptoms | interventions — Mindfulness-Based Cognitive Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Other): Mindfulness-Based Cognitive Therapy
  Interventions: Behavioral: Mindfulness-Based Cognitive Therapy for Functional Disorders
- B (No Intervention): Shared care: Treatment as usual augmented by psychiatric consultation intervention to optimise treatment in the present health care system.

INTERVENTIONS:
Behavioral: Mindfulness-Based Cognitive Therapy for Functional Disorders — Mindfulness-based cognitive therapy: A manualized program will be delivered by two instructors who are experienced cognitive therapists in eight weekly 3½-hour group training sessions and one follow-up session after a month involving up to 12 patients with somatoform disorders. The patients must be willing and able to attend and devote up to 1 hour per day for homework.
  The therapy is compared with a group of controls receiving shared care defined as: Treatment as usual augmented by psychiatric consultation intervention: The patients are offered a psychiatric consultation after the assessment interview. It is the aim to optimise treatment in the present health care system.
  Arms: A

SUMMARY:
The aim of the study is to examine the efficacy of Mindfulness-Based Cognitive Therapy (MBCT) in patients with functional disorders defined as severe Bodily Distress Disorder.

Hypothesis: MBCT can ameliorate the symptoms of FD defined as severe Bodily Distress Disorder and decrease health care utilization beyond the effect of shared care. Patients treated with MBCT will function better physically and socially than patients treated with shared care at 12 months' follow-up.

DETAILED DESCRIPTION:
Functional Disorders (FD) are conditions where patients complain of multiple medically unexplained physical symptoms. FD defy the clinical picture of any conventionally defined disease and cannot adequately be supported by clinical or para-clinical findings. The disorders are common in all medical settings, both in primary and secondary care. The conditions range from mild to severe and disabling, they are costly for society due to the patients' high health care use, and the patients' social and functional level is reduced. There is no well-established, effective pharmacological, or psychotherapeutical treatment offer today.

In randomized controlled trials, cognitive behavioural treatment has shown to be effective for selected patient groups suffering from FD. However, only a few trials have been made, especially concerning treatment of the most severe disorders.

Randomized controlled trials on Mindfulness-Based Stress Reduction (MBSR) have shown mitigation of stress, anxiety, and dysphoria in a general population sample and reduction in total mood disturbances and stress symptoms in a medical population sample. Furthermore, RCTs in Mindfulness-Based Cognitive Therapy (MBCT) have demonstrated a 50 % reduction of depression relapse for individuals, who have experienced three or more previous episodes.

We wish to examine the efficacy of MBCT in patients with functional disorders defined as severe Bodily Distress Disorder.

ELIGIBILITY:
Inclusion Criteria:

* Functional disorder defined as Bodily Distress Disorder, severe
* Moderate to severe impairment
* The disorder's functional component can easily be separated from a coexisting well-defined physical disease
* No lifetime-diagnosis of psychosis, bipolar affective disorder, or depression with psychotic symptoms
* Age 20-50 years
* Patients of Scandinavian origin, who understand, read, write, and speak Danish

Exclusion Criteria:

* No informed consent
* An acute psychiatric disorder demanding other treatment, or if the patient is suicidal
* Abuse of narcotics or alcohol or (non-prescribed) medicine
* Pregnancy

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 150 (Actual)
Dates: Start 2007-06; Primary Completion 2009-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Physical health measured by SF-36 Physical Component Summary | End of treatment, 6 and 12 months' follow-up

SECONDARY OUTCOMES:
1. Social functioning, emotional disorders, coping: Sub-scales from SF-36, WHO-DAS II, CSQ, SCL, Whiteley-7, lifestyle factors, mindfulness scales. 2. Health care use: Data from national registers. | End of treatment, 6 and 12 months' follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Per Fink, DMSc, Study Director — The Research Clinic for Functional Disorders, Aarhus University Hospital
Locations (1):
- Per Fink, Aarhus C, Denmark